CLINICAL TRIAL: NCT00847288
Title: OptiVol® Care Pathway
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OptiVol® Care Pathway
Record Dates: First submitted 2009-02-13; First posted 2009-02-19 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; Implantable Cardioverter Defibrillator (ICD); Cardiac Resynchronization Therapy with Defibrillator (CRT D); OptiVol®
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monthly Review Arm (Experimental): Patients enrolled at centers that are assigned to the monthly review arm will have their device data reviewed monthly
  Interventions: Other: Monthly Review Arm
- Quarterly Review Arm (Active Comparator): Patients enrolled at centers that are assigned to the quarterly review arm will have their device data reviewed every 3 months
  Interventions: Other: Quarterly Review Arm

INTERVENTIONS:
Other: Monthly Review Arm — Monthly review of Cardiac Compass Trends with OptiVol. This intervention is related to disease management.
  Arms: Monthly Review Arm
Other: Quarterly Review Arm — Quarterly review of Cardiac Compass Trends with OptiVol. This intervention is related to disease management.
  Arms: Quarterly Review Arm

SUMMARY:
Medtronic, Inc. is sponsoring the OptiVol® Care Pathway Study, a prospective, randomized, multi-center, post-market clinical trial in the United States. The purpose of this clinical trial is to compare monthly versus quarterly review of Cardiac Compass® Trends with OptiVol for initiation of clinical action. It is hypothesized that monthly review of Cardiac Compass Trends with OptiVol will shorten time to clinical action as compared to quarterly review.

ELIGIBILITY:
Inclusion Criteria:

* Subject (or subject's legally authorized representative) is willing and able to sign and date written consent form and Authorization for Access to and Use of Health Information
* Subject is at least 18 years of age
* Subject is willing and able to comply with Clinical Investigation Plan
* Subject is willing and able to transmit data using Medtronic CareLink® Network
* Subject has market released right atrial (RA) (if applicable), right ventricular (RV), and left ventricular (LV) (if applicable) leads and one of the following generators implanted: Concerto® CRT-D - Model C154DWK, Virtuoso® DR ICD - Model D154AWG, Virtuoso® VR ICD - Model D154VWC, Consulta™ CRT-D - Model D224TRK, Secura™ DR ICD - Model D224DRG, Secura™ VR ICD - Model D224VRC, or any future market released Medtronic generator with wireless telemetry, Cardiac Compass with OptiVol Fluid Status Monitoring, and that is supported by the Medtronic CareLink Network

Exclusion Criteria:

* Subject is enrolled in a concurrent study with the exception of a study approved by the Medtronic Clinical Trial Leader prior to enrollment
* Subject has life expectancy of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1682 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Tang, MD, Principal Investigator — Department of Cardiovascular Medicine, Cleveland Clinic
Locations (108):
- United States (108):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Anchorage, Alaska
  - Mesa, Arizona
  - Fort Smith, Arkansas
  - Little Rock, Arkansas
  - Alhambra, California
  - Berkeley, California
  - Burbank, California
  - Chula Vista, California
  - La Jolla, California
  - Larkspur, California
  - Pomona, California
  - Rancho Mirage, California
  - Riverside, California
  - San Francisco, California
  - Torrance, California
  - Boulder, Colorado
  - Colorado Springs, Colorado
  - Brandenton, Florida
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Fort Lauderdale, Florida
  - Gainesville, Florida
  - Inverness, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Miami, Florida
  - Orlando, Florida
  - Trinity, Florida
  - Augusta, Georgia
  - Columbus, Georgia
  - Chicago, Illinois
  - Kankakee, Illinois
  - Oak Lawn, Illinois
  - Rockford, Illinois
  - Bloomington, Indiana
  - Muncie, Indiana
  - Munster, Indiana
  - Terre Haute, Indiana
  - Davenport, Iowa
  - Des Moines, Iowa
  - Ashland, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Shreveport, Louisiana
  - Bangor, Maine
  - Glen Burnie, Maryland
  - Rockville, Maryland
  - Salisbury, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Grand Blanc, Michigan
  - Grand Rapids, Michigan
  - Petosky, Michigan
  - Sterling Heights, Michigan
  - Coon Rapids, Minnesota
  - Minneapolis, Minnesota
  - Saint Cloud, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - Saint Joseph, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Reno, Nevada
  - Bridgewater, New Jersey
  - Galloway, New Jersey
  - Newark, New Jersey
  - Ocean City, New Jersey
  - Voorhees Township, New Jersey
  - Buffalo, New York
  - Fayetteville, New York
  - Garden City, New York
  - Durham, North Carolina
  - Gastonia, North Carolina
  - Greensboro, North Carolina
  - Wilmington, North Carolina
  - Minot, North Dakota
  - Akron, Ohio
  - Cleveland, Ohio
  - Kettering, Ohio
  - Poland, Ohio
  - Steubenville, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Bend, Oregon
  - Doylestown, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wynnewood, Pennsylvania
  - Columbia, South Carolina
  - Greenwood, South Carolina
  - Spartanburg, South Carolina
  - West Columbia, South Carolina
  - Germantown, Tennessee
  - Johnson City, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Corpus Christi, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Lynchburg, Virginia
  - Spokane, Washington
  - Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period of OptiVol Care Pathway Study was from April 2, 2009 to March 7, 2011.
Pre-assignment Details: There were 1682 enrollments from 106 study centers. 1668 of those enrollments met the inclusion criteria for the study and thus were randomized. Fourteen did not meet the inclusion criteria and were excluded before randomization.
Period: Overall Study
Arm/Group | Monthly Review Arm | Quarterly Review Arm
Started | 841 | 827
Completed | 811 | 780
Not Completed | 30 | 47

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monthly Review Arm | Quarterly Review Arm | Total
Number analyzed (Participants) | 841 | 827 | 1668
Age Continuous [Mean (Standard Deviation); unit: years] | 68.3 (11.8) | 67.6 (11.6) | 68.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 238 | 224 | 462
  Male | 603 | 603 | 1206
Race/Ethnicity, Customized [Number; unit: participants]
  White | 749 | 621 | 1370
  Black | 53 | 98 | 151
  American Indian | 5 | 2 | 7
  Asian | 4 | 8 | 12
  Hawaiian | 2 | 2 | 4
  Hispanic | 20 | 69 | 89
  Multiple | 0 | 3 | 3
  Other | 3 | 4 | 7
  Not Available | 5 | 20 | 25
Height [Mean (Standard Deviation); unit: inches] | 68.2 (4.0) | 68.1 (4.2) | 68.1 (4.1)
Weight [Mean (Standard Deviation); unit: lbs] | 196.5 (45.9) | 196.1 (48.8) | 196.3 (47.4)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 118.6 (17.0) | 122.7 (17.1) | 120.6 (17.2)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 69.2 (10.1) | 72.4 (10.7) | 70.8 (10.5)

OUTCOME MEASURES:

1. Primary Outcome: Compare the Time to Initiation of Clinical Action Prompted by an OptiVol Threshold Crossing Between Monthly and Quarterly Review of Cardiac Compass Trends With OptiVol
Time Frame: 1 year
Population: All patients enrolled in the study, who have eligible study device, signed inform consent, signed HIPAA, and have at least one OptiVol threshold crossing post the start date, were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Monthly Review Arm | Quarterly Review Arm
Number analyzed (Participants) | 639 | 605
months | 8.9 [7.2 to 9.9] | 12.4 [12.0 to 13.1]
Statistical Analysis 1: Comparison: Monthly Review Arm vs Quarterly Review Arm; Let TM and TQ denote the median survival time to initiation of clinical action in monthly and quarterly review groups respectively. Null Hypothesis (HO): The time to initiation of clinical action is not affected by review frequency (monthly versus quarterly): TM=TQ Alternative Hypothesis (HA): The time to initiation of clinical action is affected by review frequency (monthly versus quarterly): TM≠TQ Cox proportional hazard model will be fitted to estimate the hazard ratio; Test type: Superiority or Other; p = 0.0043, Regression, Cox — Cox proportional hazard model was fitted with the group effect and other key baseline variables. The p-value for the main group effect is 0.0043, with an estimated hazard ratio of 1.5, monthly vs quarterly; Hazard Ratio (HR) = 1.5, 95% CI 2-sided [1.1 to 2.0]

2. Secondary Outcome: Compare Changes in Subject Self-care Over Time in the Monthly Review Arm vs. Quarterly Review Arm
Description: There are 3 summary scale scores for the Self-Care of Heart Failure Index (SCHFI) form: self-care maintenance score (Section A), management score (Section B), and confidence score (Section C). Each scale score is standardized to a 0 to 100 range, with 0 indicating the worst and 100 indicating the best performance for each scale score.
  Here, changes in each scale score between 6 month follow-up and baseline and between 12 month follow-up and baseline are the secondary outcome measures. Specifically, change at 6 (or 12) month follow-up is calculated as a scale score at 6 (or 12) month follow-up subtracts that at baseline. These changes range from -100 to 100 with 0 indicating no change at all, -100 indicating maximum decrease and 100 indicating maximum increase that is possible from baseline for a self-care scale score.
Time Frame: 1 year
Population: For each component, the subject needs to have baseline and 6 (or 12) month measurements to calculate the changes. Subjects included for the each component are as following:
  Maintenance (or Confidence): 720 and 675 for monthly and quarterly arms at 6 mo, respectively, 640 and 588 at 12 mo. Management, 166 and 141 at 6 mo, 166 and 104 at 12 mo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Monthly Review Arm | Quarterly Review Arm
Number analyzed (Participants) | 720 | 640
units on a scale
  Maintenance (6 mo) | 1.94 (13.31) | -0.77 (13.65)
  Management (6 mo) | -1.72 (24.33) | -1.05 (22.99)
  Confidence (6 mo) | -1.19 (20.71) | -2.46 (20.96)
  Maintenance (12 mo) | 1.1 (13.16) | -1.42 (14.73)
  Management (12 mo) | -2.32 (24.96) | -4.17 (25.27)
  Confidence (12 mo) | 0.32 (21.64) | -1.74 (22.65)

3. Secondary Outcome: Identify Patient Groups Who Are More Likely to Have Clinical Actions Triggered by Monthly Rather Than Quarterly Reviews
Description: The binary outcome of having clinical actions taken (Yes/No) is recorded within one month interval for the monthly review group, and within three months interval for the quarterly review group. To make the endpoints of both groups comparable, data from monthly review group are converted as they were collected quarterly. For example, the month 1, 2 and 3 visits of monthly review group are combined as one visit. If there is at least one action taken in any of these three monthly visits, the action taken variable for the combined visit will be recorded as 'yes'. Unscheduled visits in both groups are lumped to the next quarterly time point.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: percentage of visits with action
Units Other Than Participants: visits
Arm/Group | Monthly Review Arm | Quarterly Review Arm
Number analyzed (Participants) | 813 | 780
Number analyzed (visits) | 3065 | 2732
percentage of visits with action | 0.26 [0.24 to 0.28] | 0.19 [0.17 to 0.20]
Statistical Analysis 1: Comparison: Monthly Review Arm vs Quarterly Review Arm; The probability of action taken in three months interval is evaluated using the generalized estimating equations (GEE) method under a logistic regression model. Univariate analysis is performed first for potential predictors and only those with a p-value less than 0.10 through univariate analysis are included in the multivariate model. Here we report the odds ratio of monthly arm against quarterly arm, adjusting for OptiVol crossing, new or chronic device, and AF or no AF; Test type: Superiority or Other; p = 0.0001, logistic GEE for repeated observations; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.20 to 1.74]

4. Secondary Outcome: Compare the Time to Initiation of Clinical Action With or Without an OptiVol Threshold Crossing Between Monthly and Quarterly Review of Cardiac Compass Trends With OptiVol
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Monthly Review Arm | Quarterly Review Arm
Number analyzed (Participants) | 813 | 780
months | 9.0 [7.2 to 10.8] | 13.2 [12.6 to 16.3]

ADVERSE EVENTS:
Description: Adverse Events were not collected for this study.
Arm/Group | Monthly Review Arm | Quarterly Review Arm
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other